CLINICAL TRIAL: NCT01562171
Title: Lentils as a Functional Food to Improve Glucose Tolerance and Decrease Cardiovascular Disease Risk in Hypercholesterolemic Overweight Individuals
Brief Title: Lentils as a Functional Food to Improve Glucose and Decrease Cardiovascular Risk
Acronym: LEN-0-2012
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Glycemic Index Laboratories, Inc (Industry); Agriculture and Agri-Food Canada (Other Government); Saskatchewan Pulse Growers (Other)
Responsible Party: Principal Investigator, Dr. Carla Taylor, Professor, Department of Human Nutritional Sciences, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B2012:010
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Hypercholesterolemia
Keywords: Overweight; Obese; Obesity; Cholesterol; Hypercholesterolemia; LDL-Cholesterol
MeSH Terms: conditions — Obesity; Hypercholesterolemia; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cooked Lentils (Experimental): The study group will be asked to consume food items containing one serving of (0.3 cups) of cooked lentils per day for the first 5 days, followed by one serving of (0.6 cups) of cooked lentils per day 5 times per week (equivalent of 3 cups cooked lentils per week) for the remainder of the 12-week schedule.
  Interventions: Other: Cooked Lentils
- Potato-Based Foods (Active Comparator): The control group will be asked to consume one serving per day of potato-based foods in matrices similar to those containing lentils in the same 12-week schedule, including the smaller serving size for the first 5 days.
  Interventions: Other: Potato-Based Foods

INTERVENTIONS:
Other: Cooked Lentils — Consume food items containing one serving of (0.3 cups) of cooked lentils per day for the first 5 days, followed by one serving of (0.6 cups) of cooked lentils per day 5 times per week (equivalent of 3 cups cooked lentils per week) for the remainder of the 12-week schedule.
  Arms: Cooked Lentils
Other: Potato-Based Foods — Control - Consumption of one serving per day of potato-based foods in matrices similar to those containing lentils in the same 12-week schedule, including the smaller serving size for the first 5 days.
  Arms: Potato-Based Foods

SUMMARY:
Compared to control foods, consumption of 3 cups of cooked lentils given weekly for 12 weeks will significantly improve glucose tolerance and lower LDL-cholesterol in individuals with high cholesterol and obesity.

DETAILED DESCRIPTION:
This is a multi-site, randomized, controlled, parallel group food study designed to examine the health benefits, specifically glucose tolerance, insulin sensitivity and LDL-cholesterol in overweight individuals with a high waist circumference and elevated LDL-cholesterol. Recruitment will consist of approximately 102 overweight participants (n= 51 participants per site, at 2 sites located in Winnipeg and Toronto) with high waist circumference and elevated LDL-cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females aged 30 to 75 years;
* Body Mass Index of ≤40 kg/m2 and ≥23 kg/m2 if Asian or ≥25 kg/m2 if non-Asian;
* Waist circumference ≥94 cm for males and ≥80 cm for females of Asian ethnicity,and ≥102 cm for males and ≥88 cm of non-Asian ethnicity;
* Fasting plasma glucose <7 mmol/L;
* Fasting triglycerides <4.00 mmol/L and LDL-cholesterol >2.50 mmol/L and <5.00 mmol/L;
* Must be on a stable regime for the past 3 months if taking medications to treat hypertension or if taking vitamin and mineral/dietary/herbal supplements;
* Stable body weight (±3 kg) for the past 3 months

Exclusion Criteria:

* Previous diagnosis of type 2 diabetes;
* High pulse consumption (≥2 servings per week);
* Presence of liver disease (aspartate transaminase >2 times Upper Normal Limit), renal insufficiency (creatinine >1.5 times Upper Normal Limit); inflammatory bowel disease or other gastrointestinal disorders influencing gastrointestinal motility or nutrient absorption;
* Use of medication which influence carbohydrate metabolism (i.e., steroids), or medications used to treat diabetes or to lower blood lipids, or any active medical or surgical conditions within the past 3 months;
* Conditions or medications which are likely to increase the risk to the participants or study personnel, or to reduce the ability of the participant to comply with the protocol, or affect the results;
* History of gastrointestinal reactions or allergies to lentils or potato-based foods, or to one or more ingredients in the study foods which significantly limits the number of study foods that can be consumed.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To examine the effect of lentils on glucose tolerance and LDL-cholesterol. | 12 weeks

SECONDARY OUTCOMES:
To examine the effect of lentils on glycated hemoglobin; fasting plasma glucose, insulin, triglycerides, HDL-cholesterol and C-reactive protein. | 12 weeks

OTHER OUTCOMES:
To examine the effect of lentils on vascular responsiveness, and biomarkers of vascular function, inflammation and metabolism. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taylor, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - I.H. Asper Clinical Research Institute, Winnipeg, Manitoba
  - Glycemic Index Laboratories, Incorporated, Toronto, Ontario

REFERENCES:
- [Background] Wilson PW, D'Agostino RB, Sullivan L, Parise H, Kannel WB. Overweight and obesity as determinants of cardiovascular risk: the Framingham experience. Arch Intern Med. 2002 Sep 9;162(16):1867-72. doi: 10.1001/archinte.162.16.1867. PMID 12196085
- [Background] Calkin AC, Allen TJ. Diabetes mellitus-associated atherosclerosis: mechanisms involved and potential for pharmacological invention. Am J Cardiovasc Drugs. 2006;6(1):15-40. doi: 10.2165/00129784-200606010-00003. PMID 16489846
- [Background] Juvenile diabetes Research Foundation (2005) http://www.jdrf.org.au/publications/factsheets/complications.html Accessed July 30, 2009.
- [Background] Li TY, Rana JS, Manson JE, Willett WC, Stampfer MJ, Colditz GA, Rexrode KM, Hu FB. Obesity as compared with physical activity in predicting risk of coronary heart disease in women. Circulation. 2006 Jan 31;113(4):499-506. doi: 10.1161/CIRCULATIONAHA.105.574087. PMID 16449729
- [Background] Statistics Canada: http://www.hc-sc.gc.ca/dc-ma/diabete/index_e.html. Accessed July 30, 2009.
- [Background] Festa A, Williams K, D'Agostino R Jr, Wagenknecht LE, Haffner SM. The natural course of beta-cell function in nondiabetic and diabetic individuals: the Insulin Resistance Atherosclerosis Study. Diabetes. 2006 Apr;55(4):1114-20. doi: 10.2337/diabetes.55.04.06.db05-1100. PMID 16567536
- [Background] Lasker RD. The diabetes control and complications trial. Implications for policy and practice. N Engl J Med. 1993 Sep 30;329(14):1035-6. doi: 10.1056/NEJM199309303291410. No abstract available. PMID 8366905
- [Background] Kreisberg RA. Diabetic dyslipidemia. Am J Cardiol. 1998 Dec 17;82(12A):67U-73U; discussion 85U-86U. doi: 10.1016/s0002-9149(98)00848-0. PMID 9915665
- [Background] Wolever TM, Mehling C, Chiasson JL, Josse RG, Leiter LA, Maheux P, Rabasa-Lhoret R, Rodger NW, Ryan EA. Low glycaemic index diet and disposition index in type 2 diabetes (the Canadian trial of carbohydrates in diabetes): a randomised controlled trial. Diabetologia. 2008 Sep;51(9):1607-15. doi: 10.1007/s00125-008-1093-x. Epub 2008 Jul 22. PMID 18648764
- [Background] Sievenpiper JL, Kendall CW, Esfahani A, Wong JM, Carleton AJ, Jiang HY, Bazinet RP, Vidgen E, Jenkins DJ. Effect of non-oil-seed pulses on glycaemic control: a systematic review and meta-analysis of randomised controlled experimental trials in people with and without diabetes. Diabetologia. 2009 Aug;52(8):1479-95. doi: 10.1007/s00125-009-1395-7. Epub 2009 Jun 13. PMID 19526214
- [Background] Pulse Canada: http://www.pulsecanada.com/uploads/9f/96/9f9658890a7180395b648f83f26978c5/09-Apr-20-Clinical-Trial-release.pdf Accessed July 30, 2009.
- [Background] Rizkalla SW, Bellisle F, Slama G. Health benefits of low glycaemic index foods, such as pulses, in diabetic patients and healthy individuals. Br J Nutr. 2002 Dec;88 Suppl 3:S255-62. doi: 10.1079/BJN2002715. PMID 12498625
- [Background] Wylie-Rosett J, Segal-Isaacson CJ, Segal-Isaacson A. Carbohydrates and increases in obesity: does the type of carbohydrate make a difference? Obes Res. 2004 Nov;12 Suppl 2:124S-9S. doi: 10.1038/oby.2004.277. PMID 15601960
- [Background] Delzenne NM, Cani PD. A place for dietary fibre in the management of the metabolic syndrome. Curr Opin Clin Nutr Metab Care. 2005 Nov;8(6):636-40. doi: 10.1097/01.mco.0000171124.06408.71. PMID 16205465
- [Background] Anderson JW, Major AW. Pulses and lipaemia, short- and long-term effect: potential in the prevention of cardiovascular disease. Br J Nutr. 2002 Dec;88 Suppl 3:S263-71. doi: 10.1079/BJN2002716. PMID 12498626
- [Background] Frick M, Weidinger F. Endothelial function: a surrogate endpoint in cardiovascular studies? Curr Pharm Des. 2007;13(17):1741-50. doi: 10.2174/138161207780831211. PMID 17584104
- [Background] Tsuda T, Ueno Y, Aoki H, Koda T, Horio F, Takahashi N, Kawada T, Osawa T. Anthocyanin enhances adipocytokine secretion and adipocyte-specific gene expression in isolated rat adipocytes. Biochem Biophys Res Commun. 2004 Mar 26;316(1):149-57. doi: 10.1016/j.bbrc.2004.02.031. PMID 15003523
- [Background] Hooper L, Kroon PA, Rimm EB, Cohn JS, Harvey I, Le Cornu KA, Ryder JJ, Hall WL, Cassidy A. Flavonoids, flavonoid-rich foods, and cardiovascular risk: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2008 Jul;88(1):38-50. doi: 10.1093/ajcn/88.1.38. PMID 18614722
- [Background] Risso A, Mercuri F, Quagliaro L, Damante G, Ceriello A. Intermittent high glucose enhances apoptosis in human umbilical vein endothelial cells in culture. Am J Physiol Endocrinol Metab. 2001 Nov;281(5):E924-30. doi: 10.1152/ajpendo.2001.281.5.E924. PMID 11595647
- [Background] Abdul-Ghani MA, Matsuda M, Balas B, DeFronzo RA. Muscle and liver insulin resistance indexes derived from the oral glucose tolerance test. Diabetes Care. 2007 Jan;30(1):89-94. doi: 10.2337/dc06-1519. PMID 17192339
- [Background] Phillips DI, Clark PM, Hales CN, Osmond C. Understanding oral glucose tolerance: comparison of glucose or insulin measurements during the oral glucose tolerance test with specific measurements of insulin resistance and insulin secretion. Diabet Med. 1994 Apr;11(3):286-92. doi: 10.1111/j.1464-5491.1994.tb00273.x. PMID 8033528
- [Background] American Heart Association Nutrition Committee; Lichtenstein AH, Appel LJ, Brands M, Carnethon M, Daniels S, Franch HA, Franklin B, Kris-Etherton P, Harris WS, Howard B, Karanja N, Lefevre M, Rudel L, Sacks F, Van Horn L, Winston M, Wylie-Rosett J. Diet and lifestyle recommendations revision 2006: a scientific statement from the American Heart Association Nutrition Committee. Circulation. 2006 Jul 4;114(1):82-96. doi: 10.1161/CIRCULATIONAHA.106.176158. Epub 2006 Jun 19. PMID 16785338
- [Derived] Pauls SD, Du Y, Clair L, Winter T, Aukema HM, Taylor CG, Zahradka P. Impact of Age, Menopause, and Obesity on Oxylipins Linked to Vascular Health. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):883-897. doi: 10.1161/ATVBAHA.120.315133. Epub 2020 Dec 31. PMID 33380172
- See also: Canadian Centre for Agri-Food Research in Health & Medicine (website) — http://www.sbrc.ca/ccarm/